CLINICAL TRIAL: NCT01249664
Title: A Phase-3, Multi-center, Randomized, Double-masked, Sham-controlled Study of the Efficacy, Safety, and Tolerability of Intravitreal VEGF Trap-Eye in Subjects With Choroidal Neovascularization Secondary to Pathologic Myopia
Brief Title: VEGF Trap-Eye in Choroidal Neovascularization Secondary to Pathologic Myopia (mCNV)
Acronym: Myrror
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Therapeutic Area Head, Bayer Healthcare AG
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15170
Record Dates: First submitted 2010-11-26; First posted 2010-11-30 (Estimated); Results first posted 2014-04-01 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-04

CONDITIONS: Myopia, Pathological
Keywords: sham-controlled; pathologic myopia; mCNV; choroidal neovascularization; intravitreal injection; vision loss; macular damage
MeSH Terms: conditions — Myopia, Degenerative; Choroidal Neovascularization; Vision Disorders | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Biological: VEGF Trap-Eye (BAY86-5321)
- Arm 2 (Sham Comparator)
  Interventions: Procedure: No Drug

INTERVENTIONS:
Biological: VEGF Trap-Eye (BAY86-5321) — 1 intravitreal injection of the experimental drug, followed by monthly re-injections if needed
  Arms: Arm 1
Procedure: No Drug — Sham procedure NOT involving injection of any substance; patient´s eye is anesthetized and a syringe without needle gently pressed on the cornea
  Arms: Arm 2

SUMMARY:
VEGF Trap-Eye will be tested for safety and efficacy in patients with vision loss due to choroidal neovascularization secondary to pathologic myopia. This will be a placebo-controlled trial. 3 out of 4 patients will receive an injection of VEGF Trap-Eye into the affected eye (and repeated injections if required), and 1 out of 4 patients will receive a sham injection requiring no needle stick, but making the patient unaware of whether or not he received active treatment.

Outcome of the two treatment groups will be compared after 24 weeks. From week 24, sham patients may receive active treatment.

Total duration of the study will be 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Able to read (or, if unable to read due to visual impairment, be read to verbatim by the person administering the informed consent form or a family member) and understand the informed consent form and willing to sign the informed consent form
* Signed informed consent form. In Japan only, the informed consent form for a subject under the age of 20 years will require the co-signature of the subject's legally authorized representative.
* Men and women ≥ 18 years of age
* Myopia of greater than or equal to -6 D OR axial length of greater than or equal to 26.5 mm
* Active subfoveal or juxtafoveal (within 1 to 199 μm of the center of the fovea) CNV secondary to pathologic myopia as defined by leakage on FA
* Best-corrected visual acuity of 73 to 35 letters (ETDRS equivalent of 20/40 to 20/200) in the study eye at 4 meters
* Decrease in vision in the study eye is determined by the investigator, using his/her medical judgment, to be primarily the result of the current active mCNV
* Willing, committed, and able to return for all clinic visits and complete all study-related procedures

Exclusion Criteria:

* Only one functional eye
* Ocular media of insufficient quality to obtain fundus and OCT images in the study eye
* Greatest linear dimension (GLD) of the lesion in the study eye is greater than 12 disc areas
* Recurrent mCNV in the study eye
* Aphakia in the study eye
* History or presence of CNV with an origin other than pathologic myopia in the study eye
* Ocular inflammation or external ocular inflammation in the study eye
* Concurrent disease in the study eye that would compromise BCVA or require medical or surgical intervention during the study period
* Any ocular disorder in the study eye that, in the opinion of the investigator, may confound interpretation of the study results
* Significant scarring or atrophy in the fovea that indicates substantial irreversible vision loss in the study eye
* History of idiopathic or autoimmune-associated uveitis in either eye
* Evidence at examination of infectious blepharitis, keratitis, scleritis, or conjunctivitis in either eye or current treatment for serious systemic infection
* Vitreomacular traction or traction retinal detachment, epiretinal membrane in either eye
* Any iris neovascularization and/or vitreous hemorrhage in either eye
* Uncontrolled glaucoma, or previous filtration surgery in either eye
* Prior and concomitant treatments
* In the study eye:

  * Any prior or concomitant treatment with another investigational agent for mCNV
  * Any previous panretinal photocoagulation or subfoveal thermal laser therapy
  * Any prior treatment with photodynamic therapy
  * Cataract surgery within 3 months prior to Day 1
  * Yttrium-aluminum-garnet laser capsulotomy within 2 months prior to Day 1
  * Any other intraocular surgery within 3 months prior to Day 1
  * History of vitreoretinal surgery and/or scleral buckle surgery
* Any prior treatment with anti-VEGF agents
* Previous use of intraocular or periocular corticosteroids in either eye within 3 months prior to Day 1
* Previous assignment to treatment during this study
* Uncontrolled hypertension
* History of cerebrovascular disease or myocardial infarction within 6 months prior to Baseline/Day 1
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, may affect interpretation of the results of the study, or renders the subject at high risk from treatment complications
* Women of childbearing potential without contraception, women who intend to breastfeed during the study. All subjects (both men and women) of childbearing potential who are unwilling to use adequate birth control measures during the course of the study.
* Renal failure requiring dialysis or renal transplant
* Participation in an investigational study within 30 days prior to Screening/Visit 1 that involved treatment with any drug (excluding vitamins and minerals) or device
* Known serious allergy to the fluorescein sodium for injection in angiography or Verteporfin
* Inability to obtain fundus photographs or fluorescein angiograms of sufficient quality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2010-12; Primary Completion 2013-02 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (18):
- Kowloon, Hong Kong
- Japan (13):
  - Nagoya, Aichi-ken
  - Urayasu, Chiba
  - Matsuyama, Ehime
  - Fukuoka, Fukuoka
  - Fukushima, Fukushima
  - Kyoto, Kyoto
  - Sendai, Miyagi
  - Osaka, Osaka
  - Suita, Osaka
  - Ōtsu, Shiga
  - Bunkyo-ku, Tokyo
  - Chiyoda-ku, Tokyo
  - Shinjuku-ku, Tokyo
- Singapore, Singapore
- Seoul, South Korea
- Taiwan (2):
  - Taipei
  - Taoyuan District

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 20 study centers in 5 countries. Recruitment period: 17 Dec 2010 - 28 Feb 2013.
Pre-assignment Details: A total of 173 participants were screened.
Groups:
- Aflibercept Injection First, Then Aflibercept or Sham: Participants received a single 2 mg dose of Intravitreal Aflibercept Injection (IAI) (EYLEA, VEGF Trap-Eye, BAY86-5321) at baseline (Week 0). Following this, participants were monitored every 4 weeks and received an injection at these visits up to week 44 only if the Choroidal neovascularization (CNV) persisted or recurred, i.e. protocol defined re-treatment criteria were met. If these re-treatment criteria were not met at a given visit, participant received a sham injection.
- Sham Treatment First, Then Aflibercept Injection or Sham: Participant received a sham injection every 4 weeks from Week 0 to Week 20. At Week 24, participants received a single 2 mg Intravitreal Aflibercept Injection (IAI) (EYLEA, VEGF Trap-Eye, BAY86-5321). Following this, participants were monitored every 4 weeks and received an injection at these visits up to week 44 only if the Choroidal neovascularization (CNV) persisted or recurred, i.e. protocol defined re-treatment criteria were met. If these re-treatment criteria were not met at a given visit, participant received a sham injection.
Period: Overall Study
Arm/Group | Aflibercept Injection First, Then Aflibercept or Sham | Sham Treatment First, Then Aflibercept Injection or Sham
Started | 91 | 31
Participants Received Treatment | 91 (Safety population) | 31 (Safety population)
Fulfilled Requirements of FAS Population | 90 (Full Analysis Set (FAS) population: Basis of efficacy evaluation) | 31 (FAS population: Basis of efficacy evaluation)
Completed 24 Weeks Treatment | 83 (Withdrawal from treatment does not equal to withdrawal from study.) | 25 (Withdrawal from treatment does not equal to withdrawal from study.)
Completed 48 Weeks Treatment | 78 | 24
Completed | 85 (Completers of study visits up to week 48) | 31 (Completers of study visits up to week 48)
Not Completed | 6 | 0
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aflibercept Injection First, Then Aflibercept or Sham | Sham Treatment First, Then Aflibercept Injection or Sham | Total
Number analyzed (Participants) | 90 | 31 | 121
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.5 (13.7) | 57.5 (12.1) | 58.2 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 27 | 92
  Male | 25 | 4 | 29
Baseline Best Corrected Visual Acuity (BCVA) letter scores [Mean (Standard Deviation); unit: Letters correctly read] — Information retrieved from all baseline participants. Only participants with a ETDRS (Early Treatment Diabetic Retinopathy Study) Best Corrected Visual Acuity letter score of 73 to 35 (= Acuity of 20/40 to 20/200) in the study eye at 4 meters were included; a higher score represents better functioning.
  Letters correctly read | 56.4 (9.8) | 56.6 (8.9) | 56.5 (9.5)
Baseline Central Retinal Thickness by Optical Coherence Tomography (OCT) [Mean (Standard Deviation); unit: µm] | 349.7 (91.3) | 354.2 (107.2) | 350.9 (95.2)
Baseline intraocular pressure [Mean (Standard Deviation); unit: mm Hg] | 15.2 (2.7) | 15.8 (2.8) | 15.4 (2.7)
Number of participants by category of time since mCNV diagnosis [Number; unit: Participants]
  >= 2 months | 17 | 7 | 24
  < 2 months | 73 | 24 | 97
Baseline National Eye Institute 25-item Visual Function Questionnaire (NEI VFQ-25) total score [Mean (Standard Deviation); unit: scores on a scale] — The NEI VFQ-25 total score ranges from 0-100 with a score of 0 being the worst outcome and 100 being the best outcome. The NEI VFQ questionnaire is organized as a collection of subscales which are all scored from 0-100. To reach the overall composite score, each sub-scale score is averaged in order to give each sub-scale equal weight.
  scores on a scale | 70.47 (13.48) | 72.73 (15.29) | 71.04 (13.94)
European questionnaire 5 dimensions (EQ-5D) total score [Mean (Standard Deviation); unit: score on a scale] — The EQ-5D total score ranges from -0.594 to 1.000 with -0.594 being the worst.
  score on a scale | 0.88 (0.18) | 0.88 (0.15) | 0.88 (0.18)
Race [Number; unit: Participants]
  Asian | 90 | 31 | 121
  White | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline Choroidal neovascularization (CNV) size [Mean (Standard Deviation); unit: disc area] — Disc Area is a ophthalmological unit of measuring areas. 1 Disc area = 2.54 millimeters squared mm^2.
  disc area | 0.4086 (0.5028) | 0.3334 (0.3413) | 0.3894 (0.4666)
Baseline area of leakage [Mean (Standard Deviation); unit: disc area] — Disc Area is a ophthalmological unit of measuring areas. 1 Disc area = 2.54 millimeters squared mm^2.
  disc area | 0.7005 (0.6830) | 0.6867 (0.5563) | 0.6970 (0.6507)
Duration of disease [Mean (Standard Deviation); unit: days] | 145.6 (437.4) | 177.1 (512.0) | 153.7 (455.6)
Baseline axial length [Mean (Standard Deviation); unit: millimeter (mm)] | 28.791 (1.524) | 28.610 (1.696) | 28.745 (1.564)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Best Corrected Visual Acuity (BCVA) as Measured by Early Treatment Diabetic Retinopathy Study (ETDRS) From Baseline to Week 24 - Last Observation Carried Forward (LOCF)
Description: Defined study baseline range of ETDRS Best Corrected Visual Acuity letter score of 73 to 35 letters (ETDRS equivalent of 20/40 to 20/200) in the study eye; a higher score represents better functioning.
Time Frame: Baseline, Week 24
Measure: Mean (Standard Deviation); unit: Letters correctly read
Arm/Group | Aflibercept Injection First, Then Aflibercept or Sham | Sham Treatment First, Then Aflibercept Injection or Sham
Number analyzed (Participants) | 90 | 31
Letters correctly read | 12.1 (8.3) | -2.0 (9.7)
Statistical Analysis 1: Comparison: Aflibercept Injection First, Then Aflibercept or Sham vs Sham Treatment First, Then Aflibercept Injection or Sham; Null hypothesis was equality in change from baseline to Week 24 in BCVA total letter score between Eylea and Sham; Test type: Superiority or Other; p < 0.0001, ANCOVA — No adjustment on P value, this is for the primary efficacy analysis; ANCOVA model, including treatment groups and country (country designations) as fixed effects and baseline BCVA as a covariate; Difference in least square means = 14.1, 95% CI 2-sided [10.8 to 17.4] — The difference is calculated as Eylea minus Sham. A positive value indicates Eylea showed a higher change in BCVA total score until week 24 compared to Sham

2. Secondary Outcome: Percentage of Participants Who Gained at Least 15 Letters in BCVA as Measured by ETDRS at Week 24 Using the LOCF Approach
Description: Defined study baseline range of Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) letter score of 73 to 35 letters (ETDRS equivalent of 20/40 to 20/200) in the study eye; a higher score represents better functioning. Nominator = (Number of participants who maintained vision * 100); Denominator = Number of participants analyzed.
Time Frame: Baseline, Week 24
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept Injection First, Then Aflibercept or Sham | Sham Treatment First, Then Aflibercept Injection or Sham
Number analyzed (Participants) | 90 | 31
Percentage of participants | 38.9 | 9.7
Statistical Analysis 1: Comparison: Aflibercept Injection First, Then Aflibercept or Sham vs Sham Treatment First, Then Aflibercept Injection or Sham; Null hypothesis of difference of Eylea minus Sham of 0 was tested; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel — No adjustment on P value, since this test was only conducted formally under the primary efficacy evaluation was significant; CMH adjusted difference = 29.2, 95% CI 2-sided [14.4 to 44.0] — A two-sided Cochran-Mantel-Haenszel method at level 5% weight-adjusted by country (country designations) was used to conduct the superiority test

3. Secondary Outcome: Mean Change in Best Corrected Visual Acuity (BCVA) as Measured by ETDRS From Baseline to Week 24 - Observed Cases
Description: Data as observed at visit, no carrying forward from latest observation if missing data at later time points. Defined study baseline range of ETDRS Best Corrected Visual Acuity letter score of 73 to 35 letters (ETDRS equivalent of 20/40 to 20/200) in the study eye; a higher score represents better functioning.
Time Frame: Baseline, Week 24
Measure: Mean (Standard Deviation); unit: Letters correctly read
Arm/Group | Aflibercept Injection First, Then Aflibercept or Sham | Sham Treatment First, Then Aflibercept Injection or Sham
Number analyzed (Participants) | 84 | 25
Letters correctly read | 12.0 (8.4) | -0.8 (9.3)
Statistical Analysis 1: Comparison: Aflibercept Injection First, Then Aflibercept or Sham vs Sham Treatment First, Then Aflibercept Injection or Sham; Test type: Superiority or Other; p < 0.0001, ANCOVA; Difference in least square means = 13.1, 95% CI 2-sided [9.4 to 16.7]

4. Secondary Outcome: Percentage of Participants Who Gained at Least 10 Letters in BCVA at Week 24 - LOCF
Description: as for outcome 2
Time Frame: Baseline, Week 24
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept Injection First, Then Aflibercept or Sham | Sham Treatment First, Then Aflibercept Injection or Sham
Number analyzed (Participants) | 90 | 31
Percentage of participants | 63.3 | 12.9
Statistical Analysis 1: Comparison: Aflibercept Injection First, Then Aflibercept or Sham vs Sham Treatment First, Then Aflibercept Injection or Sham; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted difference = 50.5, 95% CI 2-sided [35.0 to 66.0]

5. Secondary Outcome: Percentage of Participants Who Gained at Least 5 Letters in BCVA at Week 24 - LOCF
Description: as for outcome 2
Time Frame: Baseline, Week 24
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept Injection First, Then Aflibercept or Sham | Sham Treatment First, Then Aflibercept Injection or Sham
Number analyzed (Participants) | 90 | 31
Percentage of participants | 83.3 | 19.4
Statistical Analysis 1: Comparison: Aflibercept Injection First, Then Aflibercept or Sham vs Sham Treatment First, Then Aflibercept Injection or Sham; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted difference = 64.0, 95% CI 2-sided [47.8 to 80.3]

6. Secondary Outcome: Percentage of Participants Who Gained at Least 15 Letters in BCVA at Week 48 - LOCF
Description: as for outcome 2
Time Frame: Baseline, Week 48
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept Injection First, Then Aflibercept or Sham | Sham Treatment First, Then Aflibercept Injection or Sham
Number analyzed (Participants) | 90 | 31
Percentage of participants | 50.0 | 29.0
Statistical Analysis 1: Comparison: Aflibercept Injection First, Then Aflibercept or Sham vs Sham Treatment First, Then Aflibercept Injection or Sham; Test type: Superiority or Other; p = 0.0308, Cochran-Mantel-Haenszel; CMH adjusted difference = 21.0, 95% CI 2-sided [1.9 to 40.1]

7. Secondary Outcome: Percentage of Participants Who Gained at Least 10 Letters in BCVA at Week 48 - LOCF
Description: as for outcome 2
Time Frame: Baseline, Week 48
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept Injection First, Then Aflibercept or Sham | Sham Treatment First, Then Aflibercept Injection or Sham
Number analyzed (Participants) | 90 | 31
Percentage of participants | 68.9 | 41.9
Statistical Analysis 1: Comparison: Aflibercept Injection First, Then Aflibercept or Sham vs Sham Treatment First, Then Aflibercept Injection or Sham; Test type: Superiority or Other; p = 0.0075, Cochran-Mantel-Haenszel; CMH adjusted difference = 27.0, 95% CI 2-sided [7.2 to 46.8]

8. Secondary Outcome: Percentage of Participants Who Gained at Least 5 Letters in BCVA at Week 48 - LOCF
Description: as for outcome 2
Time Frame: Baseline, Week 48
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept Injection First, Then Aflibercept or Sham | Sham Treatment First, Then Aflibercept Injection or Sham
Number analyzed (Participants) | 90 | 31
Percentage of participants | 87.8 | 45.2
Statistical Analysis 1: Comparison: Aflibercept Injection First, Then Aflibercept or Sham vs Sham Treatment First, Then Aflibercept Injection or Sham; Test type: Superiority or Other; p < .0001, Cochran-Mantel-Haenszel; CMH adjusted difference = 42.7, 95% CI 2-sided [23.7 to 61.6]

9. Secondary Outcome: Percentage of Participants Who Lost at Least 15 Letters in BCVA at Week 24 - LOCF
Description: as for outcome 2
Time Frame: Baseline, Week 24
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept Injection First, Then Aflibercept or Sham | Sham Treatment First, Then Aflibercept Injection or Sham
Number analyzed (Participants) | 90 | 31
Percentage of participants | 0 | 6.5
Statistical Analysis 1: Comparison: Aflibercept Injection First, Then Aflibercept or Sham vs Sham Treatment First, Then Aflibercept Injection or Sham; Test type: Superiority or Other; p = 0.1478, Cochran-Mantel-Haenszel; CMH adjusted difference = -6.5, 95% CI 2-sided [-15.2 to 2.3]

10. Secondary Outcome: Percentage of Participants Who Lost at Least 10 Letters in BCVA at Week 24 - LOCF
Description: as for outcome 2
Time Frame: Baseline, Week 24
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept Injection First, Then Aflibercept or Sham | Sham Treatment First, Then Aflibercept Injection or Sham
Number analyzed (Participants) | 90 | 31
Percentage of participants | 0 | 25.8
Statistical Analysis 1: Comparison: Aflibercept Injection First, Then Aflibercept or Sham vs Sham Treatment First, Then Aflibercept Injection or Sham; Test type: Superiority or Other; p = 0.0006, Cochran-Mantel-Haenszel; CMH adjusted difference = -25.8, 95% CI 2-sided [-40.6 to -11.0]

11. Secondary Outcome: Percentage of Participants Who Lost at Least 5 Letters in BCVA at Week 24 - LOCF
Description: as for outcome 2
Time Frame: Baseline, Week 24
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept Injection First, Then Aflibercept or Sham | Sham Treatment First, Then Aflibercept Injection or Sham
Number analyzed (Participants) | 90 | 31
Percentage of participants | 3.3 | 35.5
Statistical Analysis 1: Comparison: Aflibercept Injection First, Then Aflibercept or Sham vs Sham Treatment First, Then Aflibercept Injection or Sham; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; CMH adjusted difference = -32.2, 95% CI 2-sided [-48.1 to -16.3]

12. Secondary Outcome: Percentage of Participants Who Lost at Least 15 Letters in BCVA at Week 48 - LOCF
Description: as for outcome 2
Time Frame: Baseline, Week 48
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept Injection First, Then Aflibercept or Sham | Sham Treatment First, Then Aflibercept Injection or Sham
Number analyzed (Participants) | 90 | 31
Percentage of participants | 1.1 | 6.5
Statistical Analysis 1: Comparison: Aflibercept Injection First, Then Aflibercept or Sham vs Sham Treatment First, Then Aflibercept Injection or Sham; Test type: Superiority or Other; p = 0.2446, Cochran-Mantel-Haenszel; CMH adjusted difference = -5.3, 95% CI 2-sided [-14.4 to 3.7]

13. Secondary Outcome: Percentage of Participants Who Lost at Least 10 Letters in BCVA at Week 48 - LOCF
Description: as for outcome 2
Time Frame: Baseline, Week 48
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept Injection First, Then Aflibercept or Sham | Sham Treatment First, Then Aflibercept Injection or Sham
Number analyzed (Participants) | 90 | 31
Percentage of participants | 1.1 | 22.6
Statistical Analysis 1: Comparison: Aflibercept Injection First, Then Aflibercept or Sham vs Sham Treatment First, Then Aflibercept Injection or Sham; Test type: Superiority or Other; p = 0.0035, Cochran-Mantel-Haenszel; CMH adjusted difference = -21.5, 95% CI 2-sided [-35.9 to -7.0]

14. Secondary Outcome: Percentage of Participants Who Lost at Least 5 Letters in BCVA at Week 48 - LOCF
Description: as for outcome 2
Time Frame: Baseline, Week 48
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept Injection First, Then Aflibercept or Sham | Sham Treatment First, Then Aflibercept Injection or Sham
Number analyzed (Participants) | 90 | 31
Percentage of participants | 3.3 | 29.0
Statistical Analysis 1: Comparison: Aflibercept Injection First, Then Aflibercept or Sham vs Sham Treatment First, Then Aflibercept Injection or Sham; Test type: Superiority or Other; p = 0.0012, Cochran-Mantel-Haenszel; CMH adjusted difference = -25.7, 95% CI 2-sided [-41.3 to -10.1]

15. Secondary Outcome: Mean Change in Central Retinal Thickness (CRT) as Assessed by Optical Coherence Tomography (OCT) From Baseline to Week 24 - LOCF
Description: A negative number indicates improvement (reduced thickness).
Time Frame: Baseline, Week 24
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Aflibercept Injection First, Then Aflibercept or Sham | Sham Treatment First, Then Aflibercept Injection or Sham
Number analyzed (Participants) | 90 | 31
microns | -79.1 (83.7) | -4.2 (127.4)
Statistical Analysis 1: Comparison: Aflibercept Injection First, Then Aflibercept or Sham vs Sham Treatment First, Then Aflibercept Injection or Sham; Test type: Superiority or Other; p < 0.0001, ANCOVA; Difference in least square means = -77.9, 95% CI 2-sided [-108.9 to -46.9]

16. Secondary Outcome: Mean Change in Central Retinal Thickness (CRT) as Assessed by Optical Coherence Tomography (OCT) From Baseline to Week 48 - LOCF
Description: A negative number indicates improvement (reduced thickness).
Time Frame: Baseline, Week 48
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Aflibercept Injection First, Then Aflibercept or Sham | Sham Treatment First, Then Aflibercept Injection or Sham
Number analyzed (Participants) | 90 | 31
microns | -83.1 (85.5) | -56.7 (119.0)
Statistical Analysis 1: Comparison: Aflibercept Injection First, Then Aflibercept or Sham vs Sham Treatment First, Then Aflibercept Injection or Sham; Test type: Superiority or Other; p = 0.0650, ANCOVA; Difference in least square means = -29.3, 95% CI 2-sided [-60.4 to 1.8]

17. Secondary Outcome: Mean Change in Choroidal Neovascularization (CNV) Lesion Size as Assessed by Fluorescein Angiography (FA) From Baseline to Week 24 - LOCF
Description: CNV area values measured in square millimeters, each disc area is equivalent to 2.54 mm^2 on the retina; lower values represent better outcomes
Time Frame: Baseline, Week 24
Measure: Mean (Standard Deviation); unit: Disc areas
Arm/Group | Aflibercept Injection First, Then Aflibercept or Sham | Sham Treatment First, Then Aflibercept Injection or Sham
Number analyzed (Participants) | 90 | 31
Disc areas | -0.2233 (0.3195) | 0.3007 (0.4383)
Statistical Analysis 1: Comparison: Aflibercept Injection First, Then Aflibercept or Sham vs Sham Treatment First, Then Aflibercept Injection or Sham; Test type: Superiority or Other; p < 0.0001, ANCOVA; Difference in least square means = -0.4808, 95% CI 2-sided [-0.5990 to -0.3626]

18. Secondary Outcome: Mean Change in Choroidal Neovascularization (CNV) Lesion Size as Assessed by Fluorescein Angiography (FA) From Baseline to Week 48 - LOCF
Description: as for outcome 17
Time Frame: Baseline, Week 48
Measure: Mean (Standard Deviation); unit: Disc areas
Arm/Group | Aflibercept Injection First, Then Aflibercept or Sham | Sham Treatment First, Then Aflibercept Injection or Sham
Number analyzed (Participants) | 90 | 31
Disc areas | -0.1995 (0.4281) | -0.0111 (0.4031)
Statistical Analysis 1: Comparison: Aflibercept Injection First, Then Aflibercept or Sham vs Sham Treatment First, Then Aflibercept Injection or Sham; Test type: Superiority or Other; p = 0.0256, ANCOVA; Difference in least square means = -0.1346, 95% CI 2-sided [-0.2525 to -0.0167]

19. Secondary Outcome: Mean Change in European Five-dimensional Health Scale (EQ-5D) Score From Baseline to Week 24 - LOCF
Description: EQ-5D is a quality of life questionnaire based on a scale from -0.594 (worst) to 1.00 (best).
Time Frame: Baseline, Week 24
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Aflibercept Injection First, Then Aflibercept or Sham | Sham Treatment First, Then Aflibercept Injection or Sham
Number analyzed (Participants) | 90 | 31
Scores on a scale | 0.0187 (0.1749) | 0.0341 (0.1723)
Statistical Analysis 1: Comparison: Aflibercept Injection First, Then Aflibercept or Sham vs Sham Treatment First, Then Aflibercept Injection or Sham; Test type: Superiority or Other; p = 0.8690, ANCOVA; Difference in least square means = -0.0045, 95% CI 2-sided [-0.0579 to 0.0490]

20. Secondary Outcome: Mean Change in National Eye Institute 25-item Visual Function Questionnaire (NEI VFQ-25) Total Score From Baseline to Week 24 - LOCF
Description: The NEI VFQ-25 total score ranges from 0-100 with a score of 0 being the worst outcome and 100 being the best outcome. The NEI VFQ questionnaire is organized as a collection of subscales which are all scored from 0-100. To reach the overall composite score, each sub-scale score is averaged in order to give each sub-scale equal weight.
Time Frame: Baseline, Week 24
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Aflibercept Injection First, Then Aflibercept or Sham | Sham Treatment First, Then Aflibercept Injection or Sham
Number analyzed (Participants) | 90 | 31
Scores on a scale | 3.14 (10.21) | -2.58 (10.07)
Statistical Analysis 1: Comparison: Aflibercept Injection First, Then Aflibercept or Sham vs Sham Treatment First, Then Aflibercept Injection or Sham; Test type: Superiority or Other; p = 0.0104, ANCOVA; Difference of least square means = 5.21, 95% CI 2-sided [1.25 to 9.18]

21. Secondary Outcome: Percentage of Participants Who Were Withdrawn From Study Drug During the First 24 Weeks
Time Frame: Baseline, Week 24
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept Injection First, Then Aflibercept or Sham | Sham Treatment First, Then Aflibercept Injection or Sham
Number analyzed (Participants) | 90 | 31
Percentage of participants | 6.7 | 19.4

22. Secondary Outcome: Mean Change in Area of Leakage From Baseline at Week 24 - LOCF
Description: A negative change from baseline indicates improvement, ie, less leakage.
Time Frame: Baseline, Week 24
Measure: Mean (Standard Deviation); unit: Disc areas
Arm/Group | Aflibercept Injection First, Then Aflibercept or Sham | Sham Treatment First, Then Aflibercept Injection or Sham
Number analyzed (Participants) | 90 | 31
Disc areas | -0.4743 (0.4839) | 0.2094 (0.5088)
Statistical Analysis 1: Comparison: Aflibercept Injection First, Then Aflibercept or Sham vs Sham Treatment First, Then Aflibercept Injection or Sham; Test type: Superiority or Other; p < 0.0001, ANCOVA; Difference in least square means = -0.6648, 95% CI 2-sided [-0.8056 to -0.5239]

ADVERSE EVENTS:
Time Frame: From the first study drug injection until 30 days after the last study drug injection at the latest up to week 48.
Groups:
- Aflibercept Injection (Until Week 20): Participants received a 2 mg single dose of IAI at baseline (Week 20). Following this, participants were monitored every 4 weeks and received an injection at these visits up to week 20 only if the CNV persisted or recurred, i.e. protocol defined re-treatment criteria were met. If these re-treatment criteria were not met, participant received a sham injection. Participants were observed until week 24. Participants in the safety population were at risk.
- Sham Treatment (Until Week 20): Participants received a sham injection every 4 weeks from week 0 through week 20. Participants were observed until week 24. Participants in the safety population were at risk.
- Aflibercept Injection (Until Week 44): Participants who continued the study drug until week 20 were monitored every 4 weeks and received a single 2 mg dose IAI at these visits from week 24 through week 44 only if the CNV persisted or recurred, i.e. protocol defined re-treatment criteria were met. If these re-treatment criteria were not met, participant received a sham injection. Participants were observed from week 24 until week 48. Participants in the safety population were at risk.
- Sham Treatment Then Aflibercept Injection (Until Week 44): Participants who continued the sham treatment until week 20 were monitored every 4 weeks and received a single 2 mg dose IAI at these visits from week 24 through week 44 only if the CNV persisted or recurred, i.e. protocol defined re-treatment criteria were met. If these re-treatment were not met, participant received a sham injection. Participants were observed from Week 24 until Week 48. Participants in the safety population were at risk.
Arm/Group | Aflibercept Injection (Until Week 20) | Sham Treatment (Until Week 20) | Aflibercept Injection (Until Week 44) | Sham Treatment Then Aflibercept Injection (Until Week 44)
Serious Adverse Events (participants affected / at risk) | 3/91 | 0/31 | 4/91 | 0/31
Other Adverse Events (participants affected / at risk) | 30/91 | 8/31 | 18/91 | 8/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aflibercept Injection (Until Week 20) (N=91) | Sham Treatment (Until Week 20) (N=31) | Aflibercept Injection (Until Week 44) (N=91) | Sham Treatment Then Aflibercept Injection (Until Week 44) (N=31)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Choroidal neovascularisation (Eye disorders) | 0 | 0 | 1 | 0
Macular hole (Eye disorders) | 0 | 0 | 2 | 0
Pneumonia moraxella (Infections and infestations) | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aflibercept Injection (Until Week 20) (N=91) | Sham Treatment (Until Week 20) (N=31) | Aflibercept Injection (Until Week 44) (N=91) | Sham Treatment Then Aflibercept Injection (Until Week 44) (N=31)
Conjunctival haemorrhage (Eye disorders) | 7 | 1 | 7 | 1
Dry eye (Eye disorders) | 6 | 1 | 1 | 1
Eye pain (Eye disorders) | 6 | 1 | 2 | 1
Posterior capsule opacification (Eye disorders) | 0 | 0 | 0 | 3
Punctate keratitis (Eye disorders) | 4 | 3 | 5 | 3
Nausea (Gastrointestinal disorders) | 5 | 0 | 3 | 0
Herpes zoster (Infections and infestations) | 0 | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 9 | 2 | 9 | 2
Headache (Nervous system disorders) | 6 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other